CLINICAL TRIAL: NCT02310932
Title: Improving Mental Health Through Integration With Primary Care in Rural Karnataka
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH100311 (NIH); R01MH100311 (NIH)
Record Dates: First submitted 2014-12-02; First posted 2014-12-08 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Chronic Disease; Depression; Anxiety
Keywords: mental health; cardiovascular disease; diabetes; hypertension; high blood pressure
MeSH Terms: conditions — Chronic Disease; Depression; Anxiety Disorders; Psychological Well-Being; Cardiovascular Diseases; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Living Intervention (Experimental): The Healthy Living Intervention group will participate in an intervention designed to improve depression, anxiety, diabetes and CVD outcomes. This will be achieved through a 12 month intervention which consists of participation in healthy living groups and integrated collaborative clinic care at their Primary Health Clinic (PHC).
  Interventions: Behavioral: Healthy Living Intervention
- Enhanced Standard Care Model (Placebo Comparator): Patients in control groups will receive an "enhanced standard" care model, which includes providing referrals for mental health needs.
  Interventions: Behavioral: Healthy Living Intervention

INTERVENTIONS:
Behavioral: Healthy Living Intervention — Patients in the intervention groups will receive integrated collaborative clinic care by their physicians, a nurse case manager and consulting psychiatrists. They will also participate in 12-month community-based "Healthy Living groups," in which cognitive and behavioral strategies are used to target health promoting behaviors, such as increased activity, improved diet, adherence to medical regimens, as well as problem-solving skills, coping skills, and social support.

SUMMARY:
This cluster Randomized Controlled Trial was designed to implement and evaluate the effects of a multi-level intervention designed to integrate mental health treatment into rural primary health clinics in South India using a collaborative care model.

DETAILED DESCRIPTION:
The prevalence of chronic non-communicable diseases, including cardiovascular disease (CVD), type-2 diabetes (DM), and common mental disorders (CMD), i.e. anxiety & depression, are increasing worldwide, including in India, where patients with CMD are underserved, especially in rural areas, due to both stigma and lack of trained providers.

Treatment of patients with dual diagnoses involves special challenges and, if left untreated, mental illness can contribute to non-adherence and worsened outcomes.

Similarly, lack of staff training in India's Primary Health Centers (PHC) can result in missed diagnoses, inappropriate treatment, and increased morbidity and suffering. A growing body of research suggests that some of these challenges can be overcome by integrating treatment of patients with co-morbid diagnoses, by using "stepped" or "collaborative" care models. Such integration may also help reduce the stigma of seeking mental health services.

We plan to address this need by implementing and evaluating a multi-level integrated intervention in collaboration with 50 Primary Health Clinics (PHC) in rural Karnataka using a cluster Randomized Controlled Trial (cRCT). Our approach is based on our team's previous clinical and behavioral research in this region and builds on a decade long collaboration between St. John's Research Institute and University of California San Francisco. This study brings together an Indo-US team of scientists and government representatives with expertise in treating and studying mental health, chronic diseases, behavior change, stigma, and in conducting large clinical trials in rural India. It also builds on the work by India's National Rural Health Mission (NRHM), which recently announced that it will add tobacco control to its agenda. If successful, this intervention thus has high potential for scale-up and sustainability.

The proposed intervention is informed by a Social Ecological Paradigm that articulates the relationship between social settings and health behavior. It uses behavior change strategies guided by Cognitive Social Theory. Patients in intervention PHCs will receive integrated collaborative clinic care by their physicians, a nurse case manager and consulting psychiatrists. They will also participate in 12-month community-based "Healthy Living groups," in which cognitive and behavioral strategies are used to target health promoting behaviors, such as increased activity, improved diet, adherence to medical regimens, as well as problem-solving skills, coping skills, and social support. These groups will initially be co-facilitated by a Master's level mental health professional and a trained lay community health outreach worker (ASHA) on a weekly basis for 3 months. During the remaining 9 months, the ASHA will conduct monthly booster sessions focusing on the maintenance of the acquired health-promoting behaviors. Patients in control PHCs will receive an "enhanced standard" care model, which includes providing referrals for mental health needs.

To ensure standardization of study procedures across settings, all control PHC staff will receive basic training in established clinical protocols, plus training in the prescription of anti-depressant medication. While this may represent somewhat of an intervention, we did not consider it ethical to allow clinically depressed patients to be treated with vitamins and anxiolytics, which are currently frequently used in the PHC.

Following a brief start-up phase to adapt measures and finalize protocols, we propose to:

1. Use ASHAs to conduct community-based screening of depression, anxiety, DM and CVD risk factors during community health fairs in the catchment areas of 25 PHCs to examine a) whether this increases subsequent diagnoses in the PHC of patients with co-morbid mental health and chronic disease diagnoses and b) whether such patients are as likely to enter and remain in treatment, compared to the standard PHC-based screening.
2. Implement and evaluate the effects of providing staff training in the collaborative care model of integrated mental health (depression, anxiety) and cardiovascular disease (hypertension, diabetes, CVD) to intervention PHC staff and compare them to control PHC staff with respect to a) knowledge and clinical skills using clinical patient vignettes, and b) perceived satisfaction reported by clinic patients in intervention and control PHCs.
3. Implement and evaluate the effects of our, multi-level integrated clinic and community-based intervention for co-morbid primary care patients compared to the enhanced standard non-integrated treatment services in a cRCT with 50 participating PHC, with regard to both mental health (depression and anxiety) and physical health (diabetes and cardiovascular disease) outcomes at post intervention, 6 month and 12 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* 30 years or older;
* Diagnosed with co-morbid CMD (Depression or Anxiety Disorder) and either
* Able and willing to consent and participate in the intervention and all assessments;
* Able to speak Kannada; and
* Mentally competent to provide consent and answer to study measures and participate in intervention (MMSE score greater than 26).

Exclusion Criteria:

* Under 30 years of age;
* Patients who are not diagnosed with co-morbid CMD (Depression or Anxiety Disorder) and either hypertension, diabetes, or diagnosed ischemic heart disease;
* Not mentally competent to provide consent and answer to study measures and participate in intervention (MMSE score > 26).
* Unable to speak Kannada; and
* Participants who do not provide contact information.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2507 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
incidence of dually diagnosed participants | 1 year
  incidence of patients presenting to Primary Health Clinic (PHC) with a dual diagnosis of depression or anxiety, and diabetes or cardiovascular disease in in the standard versus enhanced screening arms.
anxiety or depression | 1 year
  levels of anxiety or depression reported by participants, depending on initial diagnosis
blood glucose control | 1 year
  for patients presenting with diabetes
blood pressure | 1 year
  for patients presenting with hypertension
cholesterol | 1 year
  for patients presenting with hypercholesterolemia

SECONDARY OUTCOMES:
medication adherence | 1 year
  adherence to medical regimen using a Visual Analog scale. Specific regimen depends on initial diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Ekstrand, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- St. John & Research Institute/St John & Medical College & Hospital, Bangalore, Karnataka, India

REFERENCES:
- [Background] Ekstrand ML, Bharat S, Ramakrishna J, Heylen E. Blame, symbolic stigma and HIV misconceptions are associated with support for coercive measures in urban India. AIDS Behav. 2012 Apr;16(3):700-10. doi: 10.1007/s10461-011-9888-z. PMID 21290175
- [Background] Ekstrand ML, Chandy S, Heylen E, Steward W, Singh G. Developing useful highly active antiretroviral therapy adherence measures for India: the Prerana study. J Acquir Immune Defic Syndr. 2010 Mar;53(3):415-6. doi: 10.1097/QAI.0b013e3181ba3e4e. No abstract available. PMID 20190588
- [Background] Steward WT, Chandy S, Singh G, Panicker ST, Osmand TA, Heylen E, Ekstrand ML. Depression is not an inevitable outcome of disclosure avoidance: HIV stigma and mental health in a cohort of HIV-infected individuals from Southern India. Psychol Health Med. 2011 Jan;16(1):74-85. doi: 10.1080/13548506.2010.521568. PMID 21218366
- [Background] Steward WT, Bharat S, Ramakrishna J, Heylen E, Ekstrand ML. Stigma is associated with delays in seeking care among HIV-infected people in India. J Int Assoc Provid AIDS Care. 2013 Mar-Apr;12(2):103-9. doi: 10.1177/1545109711432315. Epub 2012 Jan 26. PMID 22282878
- [Background] Steward WT, Herek GM, Ramakrishna J, Bharat S, Chandy S, Wrubel J, Ekstrand ML. HIV-related stigma: adapting a theoretical framework for use in India. Soc Sci Med. 2008 Oct;67(8):1225-35. doi: 10.1016/j.socscimed.2008.05.032. Epub 2008 Jul 1. PMID 18599171
- [Background] Whooley MA. Diagnosis and treatment of depression in adults with comorbid medical conditions: a 52-year-old man with depression. JAMA. 2012 May 2;307(17):1848-57. doi: 10.1001/jama.2012.3466. PMID 22550199
- [Background] Wong JM, Na B, Regan MC, Whooley MA. Hostility, health behaviors, and risk of recurrent events in patients with stable coronary heart disease: findings from the Heart and Soul Study. J Am Heart Assoc. 2013 Sep 30;2(5):e000052. doi: 10.1161/JAHA.113.000052. PMID 24080907
- [Background] Whooley MA. To screen or not to screen? Depression in patients with cardiovascular disease. J Am Coll Cardiol. 2009 Sep 1;54(10):891-3. doi: 10.1016/j.jacc.2009.05.034. PMID 19712797
- [Background] Whooley MA, de Jonge P, Vittinghoff E, Otte C, Moos R, Carney RM, Ali S, Dowray S, Na B, Feldman MD, Schiller NB, Browner WS. Depressive symptoms, health behaviors, and risk of cardiovascular events in patients with coronary heart disease. JAMA. 2008 Nov 26;300(20):2379-88. doi: 10.1001/jama.2008.711. PMID 19033588
- [Background] Whooley MA. Depression and cardiovascular disease: healing the broken-hearted. JAMA. 2006 Jun 28;295(24):2874-81. doi: 10.1001/jama.295.24.2874. PMID 16804154
- [Background] McManus D, Pipkin SS, Whooley MA. Screening for depression in patients with coronary heart disease (data from the Heart and Soul Study). Am J Cardiol. 2005 Oct 15;96(8):1076-81. doi: 10.1016/j.amjcard.2005.06.037. Epub 2005 Aug 30. PMID 16214441
- [Background] Srinivasan K, Joseph W. A study of lifetime prevalence of anxiety and depressive disorders in patients presenting with chest pain to emergency medicine. Gen Hosp Psychiatry. 2004 Nov-Dec;26(6):470-4. doi: 10.1016/j.genhosppsych.2004.06.001. PMID 15567213
- [Background] Srinivasan K. "Blues" ain't good for the heart. Indian J Psychiatry. 2011 Jul;53(3):192-4. doi: 10.4103/0019-5545.86797. No abstract available. PMID 22135434
- [Background] Srinivasan K, Isaacs AN, Villanueva E, Lucas A, Raghunath D. Medical attribution of common mental disorders in a rural Indian population. Asian J Psychiatr. 2010 Sep;3(3):142-4. doi: 10.1016/j.ajp.2010.07.008. Epub 2010 Sep 6. PMID 23051573
- [Background] Mony PK, Jayakumar S. Preparedness for tobacco control among postgraduate residents of a medical college in bangalore. Indian J Community Med. 2011 Apr;36(2):104-8. doi: 10.4103/0970-0218.84127. PMID 21976793
- [Background] Mony PK, Vaz M. A qualitative inquiry into the application of verbal autopsy for a mortality surveillance system in a rural community of southern India. World Health Popul. 2011;13(1):30-9. doi: 10.12927/whp.2011.22514. PMID 22543418
- [Derived] Salazar LJ, Hegde D, Srinivasan K, Heylen E, Ekstrand ML. Correlates of disability among primary care patients with common mental disorders and chronic medical conditions- a cross-sectional study from rural South India. Soc Psychiatry Psychiatr Epidemiol. 2025 Apr;60(4):859-868. doi: 10.1007/s00127-024-02727-w. Epub 2024 Jul 23. PMID 39044019
- [Derived] Srinivasan K, Heylen E, Johnson Pradeep R, Mony PK, Ekstrand ML. Collaborative care compared to enhanced standard treatment of depression with co-morbid medical conditions among patients from rural South India: a cluster randomized controlled trial (HOPE Study). BMC Psychiatry. 2022 Jun 13;22(1):394. doi: 10.1186/s12888-022-04000-3. PMID 35698087
- [Derived] Thomas S, Srinivasan K, Heylen E, Ekstrand ML. Correlates of social support in individuals with a diagnosis of common mental disorders and non communicable medical diseases in rural South India. Soc Psychiatry Psychiatr Epidemiol. 2021 Sep;56(9):1623-1631. doi: 10.1007/s00127-020-01997-4. Epub 2021 Jan 1. PMID 33386410
- [Derived] Srinivasan K, Mazur A, Mony PK, Whooley M, Ekstrand ML. Improving mental health through integration with primary care in rural Karnataka: study protocol of a cluster randomized control trial. BMC Fam Pract. 2018 Sep 11;19(1):158. doi: 10.1186/s12875-018-0845-z. PMID 30205830